CLINICAL TRIAL: NCT04992520
Title: Controlled Human Infection Model Challenge/Rechallenge: Shigella Flexneri 2a and S. Sonnei Cross-protective Antigens Discovery in Healthy Adults in the United States
Brief Title: Controlled Human Infection Model Challenge/Rechallenge
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PATH (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Johns Hopkins University Center for Immunization Research (CIR) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CVIA 088
Record Dates: First submitted 2021-07-28; First posted 2021-08-05 (Actual); Results first posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2024-12

CONDITIONS: Shigellosis
MeSH Terms: conditions — Dysentery, Bacillary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Group 1A: S. sonnei 53G (Experimental): Naïve participants were challenged with 1500 colony forming units (CFU) of S. sonnei strain 53G.
  Interventions: Biological: Shigella sonnei 53G
- Group 1B: S. flexneri 2a 2457T (Naive) (Experimental): At least 3 months after the challenge in Group 1A, newly recruited naïve participants were challenged with 1500 CFU of S. flexneri 2a strain 2457T.
  Interventions: Biological: Shigella flexneri 2a 2457T
- Group 1B: S. Flexneri 2a (Veteran) (Experimental): At least 3 months after challenge with S. sonnei 53G in Group 1A, participants received a 2nd challenge with 1500 CFU of S. flexneri 2a strain 2457T.
  Interventions: Biological: Shigella flexneri 2a 2457T
- Group 2A: S. Flexneri 2a (Experimental): Naïve participants were challenged with 1500 CFU of S. flexneri 2a strain 2457T.
  Interventions: Biological: Shigella flexneri 2a 2457T
- Group 2B: S. Sonnei 53G (Naive) (Experimental): At least 3 months after the challenge in Group 2A, newly recruited naïve participants were challenged with 1500 CFU of S. sonnei 53G.
  Interventions: Biological: Shigella sonnei 53G
- Group 2B: S. Sonnei 53G (Veteran) (Experimental): At least 3 months after challenge with S. flexneri 2a in Group 2A, participants received a 2nd challenge with 1500 CFU of S. sonnei 53G.
  Interventions: Biological: Shigella sonnei 53G

INTERVENTIONS:
Biological: Shigella sonnei 53G — Shigella sonnei (S. sonnei) strain 53G (Lot 1794); Mode of Administration: Delivered with sodium bicarbonate orally after a 90 minute fast.
  Arms: Group 1A: S. sonnei 53G; Group 2B: S. Sonnei 53G (Naive); Group 2B: S. Sonnei 53G (Veteran)
Biological: Shigella flexneri 2a 2457T — Shigella flexneri (S. flexneri) strain 2457T (Lot 1617); Mode of Administration: Delivered with sodium bicarbonate orally after a 90 minute fast.
  Arms: Group 1B: S. Flexneri 2a (Veteran); Group 1B: S. flexneri 2a 2457T (Naive); Group 2A: S. Flexneri 2a

SUMMARY:
The goal of this study is to better understand Shigella immunity. The study will compare the shigellosis rate in participants previously challenged with a different Shigella serotype to the attack rate in participants not previously exposed to Shigella (naive participants).

DETAILED DESCRIPTION:
This is a single-center controlled human infection model (CHIM) study designed to assess the cross-protective efficacy and markers of protection after challenge and heterologous rechallenge with Shigella strains of different serotypes in naïve healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults, male or female, aged 18 to 50 years (all inclusive) at the time of enrollment.
2. General good health, without clinically significant medical history, physical examination findings, or clinical laboratory abnormalities per judgment of Principal Investigator (PI).
3. Willingness to participate in the study after all aspects of the protocol have been explained and written informed consent obtained.
4. Completion of a training session and demonstrated comprehension of the protocol procedures and knowledge of Shigella-associated illness by passing a written examination (70% passing score).
5. Availability for the study duration, including all planned follow-up visits.
6. Female participants must have a negative pregnancy test at screening and prior to each challenge.
7. Female participants must agree to avoid pregnancy for 29 days following the last challenge dose by use of an efficacious hormonal or barrier method of birth control during the study. Abstinence is acceptable. Female participants unable to bear children must have this documented (e.g., tubal ligation or hysterectomy).
8. Willingness to refrain from participation in a study of another investigational agent for 90 days following the last challenge dose.

Exclusion Criteria:

1. Presence of a significant medical or psychiatric condition that in the opinion of the investigator precludes participation in the study. Some medical conditions that are adequately treated and stable would not preclude entry into the study.
2. Clinically significant abnormalities in screening on physical exam or screening laboratory results as determined by PI or PI in consultation with the research monitor and Sponsor.
3. Recent receipt of another investigational product (within 30 days before enrollment).
4. Positive enzyme-linked immunosorbent assay (ELISA) and confirmatory tests for human immunodeficiency virus (HIV).
5. Positive hepatitis C (HCV) ELISA and confirmatory test (e.g., HCV ribonucleic acid (RNA)).
6. Positive hepatitis B virus surface antigen (HBsAg) by ELISA.
7. Use of any medication that affects immune function (e.g., corticosteroids and others) within 30 days preceding the first challenge or planned use during the active study period (topical and ophthalmologic steroids are allowable).
8. Evidence of impaired immune function or immune compromise (known immunodeficiency syndrome; either congenital, acquired, or iatrogenic; active autoimmune disease; repeated serious infections without known cause).
9. Immunoglobulin A (IgA) deficiency (serum IgA < 7 mg/dL or below the limit of detection of the assay).
10. Positive blood test for human leukocyte antigen (HLA)-B27.
11. Personal or family history of an inflammatory arthritis.
12. Currently pregnant or nursing.
13. Have household contacts who are < 2 years old or > 80 years old or infirm or immunocompromised.
14. Employment as a health care worker with direct patient care, in a daycare center (for children or the elderly), or direct food handler; includes individuals who work directly with food in commercial establishments.
15. Evidence of current alcohol or drug dependence, or history of dependence in the last 6 months.
16. Recent vaccination (including licensed vaccines) or receipt of an investigational product (within 30 days before challenge through 90 days following the last challenge dose). Annual influenza vaccine, an emergency authorized or licensed COVID-19 vaccine, or a TdaP or Travelers' diarrhea (TD) booster may be administered beyond 30 days after each challenge.
17. Treatment with immunoglobulins or blood products within 3 months of challenge.
18. Current or prior history of inflammatory bowel disease or irritable bowel syndrome or abnormal stool pattern (> 3/day or < 3/ week, or loose or liquid stools).
19. Chronic use of anti-diarrheal, anti-constipation, or antacid therapy; or use of these medications in the 7 days prior to challenge.
20. Use of proton pump inhibitors or H2 blockers (H2-receptor antagonists) within 48 hours prior to challenge.
21. Use of antibiotics within 7 days prior to challenge.
22. Known allergy to any 2 of the following antibiotics: ciprofloxacin, trimethoprim-sulfamethoxazole, or penicillin.
23. Symptoms of travelers' diarrhea associated with travel to countries where Shigella or other enteric infections are endemic (most of the developing world) within 3 years prior to challenge OR planned travel to endemic countries during the active study period.
24. History of shigellosis, Shigella vaccination or challenge, or a laboratory worker with known exposure to Shigella within the last 5 years.
25. Serum immunoglobulin G (IgG) titer > 2500 to either Shigella flexneri 2a or Shigella sonnei lipopolysaccharide.
26. Any other criteria which, in the investigator's opinion, would compromise the ability of the volunteer to participate in the study, the safety of the study, or the results of the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2022-04-26 (Actual); Primary Completion 2023-08-29 (Actual); Study Completion 2023-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kawsar Talaat, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Center for Immunization Research (CIR) at Johns Hopkins School of Public Health (JHSPH), Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a single-center controlled human infection model (CHIM) study conducted at the Center for Immunization Research (CIR), Johns Hopkins Bloomberg School of Public Health in Baltimore, Maryland. Healthy volunteers not previously exposed to Shigella ("Naive") were recruited for the study; once informed consent was obtained, participants were admitted to the inpatient unit at CIR for Shigella challenge and subsequent rechallenge with a different Shigella strain.
Pre-assignment Details: Naive participants were challenged with either Shigella sonnei strain 53G (Group 1A) or Shigella flexneri 2a strain 2457T (Group 2A). Approximately 3 months later, participants who continued to meet eligibility criteria received a 2nd challenge with the other Shigella strain ("Veterans"). Additional naive volunteers were enrolled alongside the veteran participants receiving their 2nd challenge; both received the same challenge agent to allow a comparison of shigellosis rates across the groups.
Groups:
- Group 1A: S. Sonnei 53G: Naïve participants were challenged with 1500 colony forming units (CFU) of Shigella sonnei (S. sonnei) strain 53G.
- Group 1B: S. Flexneri 2a (Naive): At least 3 months after the challenge in Group 1A, newly recruited naïve participants were challenged with 1500 CFU of Shigella flexneri (S. flexneri) 2a strain 2457T.
Period: Part A: First Challenge
Arm/Group | Group 1A: S. Sonnei 53G | Group 1B: S. Flexneri 2a (Naive) | Group 1B: S. Flexneri 2a (Veteran) | Group 2A: S. Flexneri 2a | Group 2B: S. Sonnei 53G (Naive) | Group 2B: S. Sonnei 53G (Veteran)
Started | 22 | 0 | 0 | 13 | 0 | 0
Completed | 21 | 0 | 0 | 11 | 0 | 0
Not Completed | 1 | 0 | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Non-compliance | 0 | 0 | 0 | 1 | 0 | 0
Period: Part B: 3 Months Later/Second Challenge
Arm/Group | Group 1A: S. Sonnei 53G | Group 1B: S. Flexneri 2a (Naive) | Group 1B: S. Flexneri 2a (Veteran) | Group 2A: S. Flexneri 2a | Group 2B: S. Sonnei 53G (Naive) | Group 2B: S. Sonnei 53G (Veteran)
Started | 0 | 5 (Newly enrolled participants received one challenge dose at the same time veteran participants received their 2nd challenge.) | 19 (Only participants who met eligibility criteria after the first challenge were eligible to receive the 2nd challenge.) | 0 | 6 (Newly enrolled participants received one challenge dose at the same time veteran participants received their 2nd challenge.) | 10 (Only participants who met eligibility criteria after the first challenge were eligible to receive the 2nd challenge.)
Completed | 0 | 5 | 17 | 0 | 6 | 9
Not Completed | 0 | 0 | 2 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline data for veteran participants who received a 2nd challenge (Groups 1B and 2B Veterans) are included in the relevant first challenge reporting group (1A or 2A).
Groups:
- Group 1A: S. Sonnei 53G: Naïve participants were challenged with 1500 CFU of S. sonnei strain 53G.
- Group 1B: S. Flexneri 2a (Naive): At least 3 months after the challenge in Group 1A, newly recruited naïve participants were challenged with 1500 CFU of S. flexneri 2a strain 2457T.
- Total: Total of all reporting groups
Arm/Group | Group 1A: S. Sonnei 53G | Group 1B: S. Flexneri 2a (Naive) | Group 1B: S. Flexneri 2a (Veteran) | Group 2A: S. Flexneri 2a | Group 2B: S. Sonnei 53G (Naive) | Group 2B: S. Sonnei 53G (Veteran) | Total
Number analyzed (Participants) | 22 | 5 | 0 | 13 | 6 | 0 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.41 (7.98) | 37.20 (7.76) |  | 34.92 (11.77) | 32.67 (7.58) |  | 35.59 (8.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 |  | 3 | 2 |  | 10
  Male | 18 | 4 |  | 10 | 4 |  | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 |  | 0 | 1 |  | 2
  Not Hispanic or Latino | 21 | 5 |  | 13 | 5 |  | 44
  Unknown or Not Reported | 0 | 0 |  | 0 | 0 |  | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 18 | 3 |  | 11 | 2 |  | 34
  White | 2 | 2 |  | 2 | 2 |  | 8
  Multiple | 1 | 0 |  | 0 | 2 |  | 3
  Unknown | 1 | 0 |  | 0 | 0 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Shigellosis Following Shigella Challenge
Description: Shigellosis was defined as:
  * Severe diarrhea: ≥ 6 loose (grade 3-5) stools within 24 hours or >800 - 999 g loose stools within any 24-hour window, or
  * Moderate diarrhea (4 - 5 loose stools within 24 hours or 401-800 g loose stools within any 24-hour window) with fever (oral temperature of ≥ 101.2°F / 38°C) OR with ≥ 1 moderate constitutional or enteric symptom OR ≥ 2 episodes of vomiting in a 24-hour period, or
  * Dysentery: ≥ 2 loose stools with gross blood (hemoccult positive) in 24 hours AND fever OR ≥ 1 moderate constitutional/enteric symptom OR ≥ 2 episodes of vomiting in 24 hours.
  Constitutional/Enteric symptoms include nausea, abdominal cramps/pain, myalgia, arthralgia, or malaise.
  Stools were graded on the following scale:
  * Grade 1, firm formed;
  * Grade 2, soft formed;
  * Grade 3, viscous opaque liquid or semi-liquid;
  * Grade 4, watery opaque liquid;
  * Grade 5, clear watery or mucoid liquid. Outcome data were evaluated by an independent, blinded adjudication board.
Time Frame: 8 days after challenge administration (Days 1-8 and Days 90-97 for challenge 2)
Population: Per-Protocol Population included participants who received the challenge dose and had no major protocol violations that were determined to potentially interfere with the clinical assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1A: S. Sonnei 53G | Group 1B: S. Flexneri 2a (Naive) | Group 1B: S. Flexneri 2a (Veteran) | Group 2A: S. Flexneri 2a | Group 2B: S. Sonnei 53G (Naive) | Group 2B: S. Sonnei 53G (Veteran)
Number analyzed (Participants) | 22 | 5 | 19 | 12 | 6 | 10
percentage of participants | 59.1 [36.4 to 79.3] | 80.0 [28.4 to 99.5] | 15.8 [3.4 to 39.6] | 58.3 [27.7 to 84.8] | 83.3 [35.9 to 99.6] | 50.0 [18.7 to 81.3]

2. Secondary Outcome: Maximum Volume of Loose Stools in Any 24-hour Period
Description: During the 8-day inpatient period after each challenge all stools were weighed and graded according to the following scale:
  * Grade 1, firm formed;
  * Grade 2, soft formed;
  * Grade 3, viscous opaque liquid or semi-liquid;
  * Grade 4, watery opaque liquid;
  * Grade 5, clear watery or mucoid liquid.
Time Frame: 8 days after challenge administration (Days 1-8 and Days 90-97 for challenge 2)
Population: Per Protocol Population
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Group 1A: S. Sonnei 53G | Group 1B: S. Flexneri 2a (Naive) | Group 1B: S. Flexneri 2a (Veteran) | Group 2A: S. Flexneri 2a | Group 2B: S. Sonnei 53G (Naive) | Group 2B: S. Sonnei 53G (Veteran)
Number analyzed (Participants) | 22 | 5 | 19 | 12 | 6 | 10
grams | 446.86 (383.47) | 656.80 (450.93) | 225.32 (285.73) | 459.67 (530.36) | 824.33 (852.98) | 294.30 (286.32)

3. Secondary Outcome: Percentage of Participants With Severe Diarrhea
Description: During the 8-day inpatient period after each challenge all stools were weighed and graded according to the following scale:
  * Grade 1, firm formed;
  * Grade 2, soft formed;
  * Grade 3, viscous opaque liquid or semi-liquid;
  * Grade 4, watery opaque liquid;
  * Grade 5, clear watery or mucoid liquid.
  Severe diarrhea was defined as ≥ 6 loose (Grade 3-5) stools within 24 hours or > 800 grams of loose (Grade 3-5) stools within any 24-hour window.
Time Frame: 8 days after challenge administration (Days 1-8 and Days 90-97 for challenge 2)
Population: Per Protocol Population
Measure: Number; unit: percentage of participants
Arm/Group | Group 1A: S. Sonnei 53G | Group 1B: S. Flexneri 2a (Naive) | Group 1B: S. Flexneri 2a (Veteran) | Group 2A: S. Flexneri 2a | Group 2B: S. Sonnei 53G (Naive) | Group 2B: S. Sonnei 53G (Veteran)
Number analyzed (Participants) | 22 | 5 | 19 | 12 | 6 | 10
percentage of participants | 50.0 | 40.0 | 10.5 | 25.0 | 50.0 | 30.0

4. Secondary Outcome: Percentage of Participants With Diarrhea of Any Severity
Description: During the 8-day inpatient period after each challenge all stools were weighed and graded according to the following scale:
  * Grade 1, firm formed;
  * Grade 2, soft formed;
  * Grade 3, viscous opaque liquid or semi-liquid;
  * Grade 4, watery opaque liquid;
  * Grade 5, clear watery or mucoid liquid.
  Participants met the criteria for diarrhea if they had ≥ 2 loose (Grade 3-5) stools weighing ≥ 200 grams within any 48-hour window or any loose stools weighing ≥ 300 grams.
Time Frame: 8 days after challenge administration (Days 1-8 and Days 90-97 for challenge 2)
Population: Per Protocol Population
Measure: Number; unit: percentage of participants
Arm/Group | Group 1A: S. Sonnei 53G | Group 1B: S. Flexneri 2a (Naive) | Group 1B: S. Flexneri 2a (Veteran) | Group 2A: S. Flexneri 2a | Group 2B: S. Sonnei 53G (Naive) | Group 2B: S. Sonnei 53G (Veteran)
Number analyzed (Participants) | 22 | 5 | 19 | 12 | 6 | 10
percentage of participants | 77.3 | 80.0 | 42.1 | 66.7 | 83.3 | 60.0

5. Secondary Outcome: Total Weight of Grade 3-5 Stools Per Participant After Challenge
Description: as for outcome 2
Time Frame: 8 days after challenge administration (Days 1-8 and Days 90-97 for challenge 2)
Population: Per Protocol Population
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Group 1A: S. Sonnei 53G | Group 1B: S. Flexneri 2a (Naive) | Group 1B: S. Flexneri 2a (Veteran) | Group 2A: S. Flexneri 2a | Group 2B: S. Sonnei 53G (Naive) | Group 2B: S. Sonnei 53G (Veteran)
Number analyzed (Participants) | 22 | 5 | 19 | 12 | 6 | 10
grams | 768.95 (741.61) | 884.40 (531.71) | 352.74 (479.56) | 747.58 (692.05) | 979.50 (1008.34) | 402.40 (403.44)

6. Secondary Outcome: Percentage of Participants With Nausea, Vomiting, Anorexia, Abdominal Pain/Cramps Rated as Moderate to Severe
Description: During the 8-day inpatient period after each challenge, nausea, vomiting, anorexia, and abdominal pain/cramps were monitored and graded (except for vomiting) according to the following:
  Mild: Discomfort noted, but no disruption of normal daily activities; slightly bothersome; relieved with or without symptomatic treatment.
  Moderate: Discomfort sufficient to reduce or affect normal daily activity to some degree; bothersome; interferes with activities, only partially relieved with symptomatic treatment.
  Severe: Discomfort sufficient to reduce or affect normal daily activity considerably; prevents regular activities; not relieved with symptomatic treatment.
  Vomiting was graded according the the following:
  Mild: One episode within a 24-hour period Moderate: Two episodes within a 24-hour period Severe: Three or more episodes within a 24-hour period.
Time Frame: 8 days after challenge administration (Days 1-8 and Days 90-97 for challenge 2)
Population: Per Protocol Population
Measure: Number; unit: percentage of participants
Arm/Group | Group 1A: S. Sonnei 53G | Group 1B: S. Flexneri 2a (Naive) | Group 1B: S. Flexneri 2a (Veteran) | Group 2A: S. Flexneri 2a | Group 2B: S. Sonnei 53G (Naive) | Group 2B: S. Sonnei 53G (Veteran)
Number analyzed (Participants) | 22 | 5 | 19 | 12 | 6 | 10
percentage of participants
  Moderate/Severe Nausea | 18.2 | 0.0 | 10.5 | 58.3 | 16.7 | 40.0
  Moderate/Severe Vomiting | 9.1 | 0.0 | 5.3 | 16.7 | 0.0 | 20.0
  Moderate/Severe Anorexia | 13.6 | 0.0 | 15.8 | 66.7 | 66.7 | 70.0
  Moderate/Severe Abdominal Pain/Cramps | 22.7 | 0.0 | 21.1 | 41.7 | 50.0 | 50.0

7. Secondary Outcome: Percentage of Participants With Dysentery
Description: During the 8-day inpatient period after each challenge all stools were weighed and graded according to the following scale:
  * Grade 1, firm formed;
  * Grade 2, soft formed;
  * Grade 3, viscous opaque liquid or semi-liquid;
  * Grade 4, watery opaque liquid;
  * Grade 5, clear watery or mucoid liquid.
  Dysentery was defined as ≥ 2 loose stools (Grade 3-5) with gross blood (hemoccult positive) in 24 hours AND fever OR ≥ 1 moderate constitutional/enteric symptom OR ≥2 episodes of vomiting in 24 hours.
  Constitutional/enteric symptoms included nausea, abdominal cramps/pain, myalgia, arthralgia, and malaise.
Time Frame: 8 days after challenge administration (Days 1-8 and Days 90-97 for challenge 2)
Population: Per Protocol Population
Measure: Number; unit: percentage of participants
Arm/Group | Group 1A: S. Sonnei 53G | Group 1B: S. Flexneri 2a (Naive) | Group 1B: S. Flexneri 2a (Veteran) | Group 2A: S. Flexneri 2a | Group 2B: S. Sonnei 53G (Naive) | Group 2B: S. Sonnei 53G (Veteran)
Number analyzed (Participants) | 22 | 5 | 19 | 12 | 6 | 10
percentage of participants | 40.9 | 20.0 | 10.5 | 41.7 | 33.3 | 60.0

8. Secondary Outcome: Time to Onset of Diarrhea
Time Frame: From challenge administration to the end of the 8-day inpatient period (Days 1-8 and Days 90-97 for challenge 2)
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Group 1A: S. Sonnei 53G | Group 1B: S. Flexneri 2a (Naive) | Group 1B: S. Flexneri 2a (Veteran) | Group 2A: S. Flexneri 2a | Group 2B: S. Sonnei 53G (Naive) | Group 2B: S. Sonnei 53G (Veteran)
Number analyzed (Participants) | 22 | 5 | 19 | 12 | 6 | 10
hours | 62.45 (28.75) | 53.95 (19.50) | 78.22 (42.16) | 53.47 (35.25) | 60.34 (24.23) | 47.46 (22.31)

9. Secondary Outcome: Number of Participants With More Severe Diarrhea
Description: During the 8-day inpatient period after each challenge all stools were weighed and graded according to the following scale:
  * Grade 1, firm formed;
  * Grade 2, soft formed;
  * Grade 3, viscous opaque liquid or semi-liquid;
  * Grade 4, watery opaque liquid;
  * Grade 5, clear watery or mucoid liquid.
  More severe diarrhea was defined as ≥ 10 loose (Grade 3-5) stools within 24 hours or ≥ 1000 grams loose stools within any 24-hour window.
Time Frame: 8 days after challenge administration (Days 1-8 and Days 90-97 for challenge 2)
Population: Per Protocol Population
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1A: S. Sonnei 53G | Group 1B: S. Flexneri 2a (Naive) | Group 1B: S. Flexneri 2a (Veteran) | Group 2A: S. Flexneri 2a | Group 2B: S. Sonnei 53G (Naive) | Group 2B: S. Sonnei 53G (Veteran)
Number analyzed (Participants) | 22 | 5 | 19 | 12 | 6 | 10
Participants | 2 | 2 | 1 | 2 | 2 | 1

10. Secondary Outcome: Number of Participants With Fever After Challenge
Description: Fever: measured oral temperature ≥ 38°C confirmed within about 20 minutes.
Time Frame: 8 days after challenge administration (Days 1-8 and Days 90-97 for challenge 2)
Population: Per Protocol Population
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1A: S. Sonnei 53G | Group 1B: S. Flexneri 2a (Naive) | Group 1B: S. Flexneri 2a (Veteran) | Group 2A: S. Flexneri 2a | Group 2B: S. Sonnei 53G (Naive) | Group 2B: S. Sonnei 53G (Veteran)
Number analyzed (Participants) | 22 | 5 | 19 | 12 | 6 | 10
Participants | 11 | 3 | 2 | 6 | 2 | 4

11. Secondary Outcome: Shigella Clinical Severity Score
Description: The Shigella clinical severity score is a composite, ordinal disease score that consists of three parameters: self-reported symptoms (arthralgia, nausea, myalgia, headache, anorexia, and abdominal cramps and pain), clinical signs (blood in stool, fever, and vomiting) and stool output (maximum loose stool output / 24 hours). Each parameter is scored based off maximum severity clinical signs, self-reported symptoms and stool output experienced over over the 8-day period.
  The Shigella clinical severity score ranges from 0 to 9, where 0 = no or mild symptoms only and 9 = severe symptoms.
Time Frame: 8 days after challenge administration (Days 1-8 and Days 90-97 for challenge 2)
Population: Per Protocol Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1A: S. Sonnei 53G | Group 1B: S. Flexneri 2a (Naive) | Group 1B: S. Flexneri 2a (Veteran) | Group 2A: S. Flexneri 2a | Group 2B: S. Sonnei 53G (Naive) | Group 2B: S. Sonnei 53G (Veteran)
Number analyzed (Participants) | 22 | 5 | 19 | 12 | 6 | 10
score on a scale | 2.95 (2.38) | 3.00 (2.55) | 1.47 (1.74) | 4.00 (2.70) | 3.50 (2.66) | 3.90 (2.64)

12. Secondary Outcome: Number of Colony Forming Units (CFUs) of the Challenge Strain Per Gram of Stool
Description: Analysis of stool samples to quantify challenge strains in the stool are not yet complete. Data will be reported once the assays have been completed.
Time Frame: 8 days after challenge administration (Days 1-8 and Days 90-97 for challenge 2)
Reporting Status: Not Posted, anticipated posting 2025-09

ADVERSE EVENTS:
Time Frame: Serious adverse events were collected up to 180 days after last challenge (a total of 270 days for participants who received 2 challenge doses). Non-serious adverse events were collected for up to 28 days after each challenge (Days 1-28 and approximate Days 90-118).
Arm/Group | Group 1A: S. Sonnei 53G | Group 1B: S. Flexneri 2a (Naive) | Group 1B: S. Flexneri 2a (Veteran) | Group 2A: S. Flexneri 2a | Group 2B: S. Sonnei 53G (Naive) | Group 2B: S. Sonnei 53G (Veteran)
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/5 | 0/19 | 0/13 | 0/6 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/5 | 0/19 | 0/13 | 0/6 | 0/10
Other Adverse Events (participants affected / at risk) | 22/22 | 5/5 | 19/19 | 10/13 | 5/6 | 9/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1A: S. Sonnei 53G (N=22) | Group 1B: S. Flexneri 2a (Naive) (N=5) | Group 1B: S. Flexneri 2a (Veteran) (N=19) | Group 2A: S. Flexneri 2a (N=13) | Group 2B: S. Sonnei 53G (Naive) (N=6) | Group 2B: S. Sonnei 53G (Veteran) (N=10)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 11 | 3 | 5 | 5 | 4 | 4
Eye pain (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 6 | 0 | 1 | 3 | 3 | 3
Abdominal pain (Gastrointestinal disorders) | 14 | 0 | 7 | 5 | 3 | 6
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal tenderness (Gastrointestinal disorders) | 4 | 0 | 2 | 2 | 3 | 1
Aphthous ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 4 | 1 | 0 | 0 | 0 | 1
Defaecation urgency (Gastrointestinal disorders) | 11 | 3 | 4 | 5 | 4 | 4
Diarrhoea (Gastrointestinal disorders) | 17 | 4 | 9 | 8 | 5 | 6
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Eructation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 9 | 0 | 6 | 6 | 4 | 4
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 11 | 1 | 2 | 3 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 7 | 0 | 3 | 7 | 4 | 4
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rectal tenesmus (Gastrointestinal disorders) | 3 | 1 | 2 | 0 | 1 | 2
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0 | 2 | 4 | 1 | 2
Chills (General disorders) | 9 | 1 | 4 | 5 | 4 | 4
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 0 | 1
Malaise (General disorders) | 10 | 3 | 4 | 7 | 5 | 6
Pyrexia (General disorders) | 11 | 3 | 2 | 6 | 2 | 4
COVID-19 (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0
Dysentery (Infections and infestations) | 9 | 1 | 2 | 5 | 2 | 6
Fungal foot infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Burns second degree (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood pressure increased (Investigations) | 4 | 2 | 4 | 2 | 0 | 1
Blood pressure systolic increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 1 | 1 | 0 | 1
Orthostatic heart rate response increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 14 | 3 | 3 | 8 | 5 | 7
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 0 | 1 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 2 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 2 | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 0 | 0 | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 1 | 3 | 7 | 3 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 8 | 0 | 2 | 7 | 3 | 3
Headache (Nervous system disorders) | 12 | 3 | 6 | 8 | 5 | 6
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 3 | 0 | 0 | 0 | 0 | 0
Paranoia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 | 0 | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 2 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-01-16): https://cdn.clinicaltrials.gov/large-docs/20/NCT04992520/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-04): https://cdn.clinicaltrials.gov/large-docs/20/NCT04992520/SAP_001.pdf